CLINICAL TRIAL: NCT02891564
Title: Computerized Intervention Targeting Cognitive Control Deficits in Depressed Adults
Brief Title: ESTIA: Computerized Intervention Targeting Cognitive Control Deficits in Depressed Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Weill Medical College of Cornell University (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Pat Arean, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001809
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Major Depression
Keywords: therapeutic video games, mobile interventions
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (R 33) (Placebo Comparator): a mobile 3D video game to be used as placebo.
  Interventions: Other: Control Mobile 3D video game
- Intervention Arm (R 33) (Experimental): a mobile 3D video game (Band Together) that has been shown to reduce older adults' susceptibility to interference by augmenting sustained attention and working memory abilities (e.g. cognitive control) through targeted adaptive algorithms.
  Interventions: Behavioral: Band Together

INTERVENTIONS:
Behavioral: Band Together — a mobile 3D video game that has been shown to reduce older adults' susceptibility to interference by augmenting sustained attention and working memory abilities (e.g. cognitive control) through targeted adaptive algorithms. This game is analogous to Project: EVO.
  Arms: Intervention Arm (R 33)
Other: Control Mobile 3D video game — expectancy-matched control game
  Arms: Control Arm (R 33)

SUMMARY:
Project:EVO is a video-game based intervention that targets neural networks associated with cognitive control. The same networks have been implicated in poor treatment response in middle and older aged adults suffering from major depression. Related work has demonstrated that healthy older adults show significant improvement in cognitive control. In a very small sample of older adults suffering from depression (n=12), we found similar improvements in selective attention and working memory after 4 weeks of intervention, along with improvements in mood comparable to participants receiving an evidence-based psychotherapy. The intent of this proposal is to first determine if at least 2/3 of participants who use Project:EVO for four weeks demonstrate significant improvements in the function of these neural networks, and if improvements are observed, to conduct a second study to see if changes in neural network functions are associated with changes in mood. If we show that Project:EVO improves neural function and mood to a greater degree than a placebo cognitive training game, we will be in a position to move onto the next phase of study, which is to demonstrate the intervention's efficacy in a much larger sample of adults with depression.

DETAILED DESCRIPTION:
Project: EVO (or "EVO") is a mobile 3D video game that has been shown to reduce older adults' susceptibility to interference by augmenting sustained attention and working memory abilities (e.g. cognitive control) through targeted adaptive algorithms. The combination of peer-reviewed validity, adaptivity, and fun video game mechanics elevates the EVO platform beyond other at-home training tools while reducing burden associated with tedious task replication. We propose to study EVO as a potential intervention for the treatment of depression, a disorder that worsens medical outcomes, promotes disability, increases expense, and complicates medical care by clouding the clinical picture and undermining treatment adherence.

R61 Phase (COMPLETE):

In this first phase, we conducted a 2-year proof of concept study to determine if EVO could engage the cognitive control network (CCN) in 30 middle-aged and older adults with major depression. Primary aims for this phase of the proposed project were to determine if EVO will result in greater CCN engagement using three levels of analysis (circuitry, performance, self-report). At the circuitry level, we measured CCN engagement by probing the system using task-based fMRI. We hypothesized that activation and functional connectivity (FC) of anterior aspects of the CCN will increase from baseline to 4-weeks after treatment initiation. Our decision to move to the next phase of the planned study was that 66% of our sample showed significant increases in CCN functions at the circuitry level of analysis (CCN activation and FC) and at either the performance level or self-report level of analysis.

R33 Phase (CURRENT):

Successful proof of concept has initiated the second phase of the ESTIA study. In this phase, we plan to conduct a 3-year pilot study to compare "Band Together" (an EVO analog) to an expectancy-matched control game in terms of CCN target engagement at the circuitry (task-based fMRI) and behavioral levels (task performance, self-report) in 60 middle-aged and older adults with major depression. In addition, we well determine if changes in target engagement are associated with changes in mood and mood-induced disability. The decision to move onto development of a proposal to study the clinical efficacy of Band Together in a larger randomized clinical trial will be based on whether we find (1) that Band Together out-performs our control condition in terms of the engagement of CCN at the circuitry and behavioral levels (2) significant associations between changes in engagement of the CCN and changes in mood and (3) that the study methods are feasible to complete (sampling rate, retention, intervention adherence, intervention acceptability and expectancy-match for our control condition).

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 45 to 75; (2) unipolar, nonpsychotic major depression (by SCID, DSM-V), (3) Hamilton Depression Rating Scale > 20; (4) off antidepressants or have been on a stable dose for 12 weeks and do not intend to change dose in the next 5 weeks, (5) capacity to consent; (6) ability to participate in MRI.

Exclusion Criteria:

* 1) Intent or plan to attempt suicide in the near future; 2) history or presence of psychiatric diagnoses other than unipolar, non-psychotic major depression or generalized anxiety disorder; 3) use of psychotropic drugs or cholinesterase inhibitors other than mild doses of benzodiazepines 4) dementia or MCI (please see Human Subjects). Participants with an MMSE score falling 1 SD below the mean score for their age and education will be excluded as well.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
CCN Function (Circuitry and Performance) | 8 weeks
  - Assess pre-post treatment change in activation (percent signal Δ) during the stroop/flanker test
CCN Function (Self-Report- Disability) | 8 weeks
  - Pre-post self-report assessment of disability via WHO Disability Assessment Scale (36-item)
CCN Function (Self-Report- Depressive Symptoms) | 8 weeks
  - Pre-post self-report assessment of depressive symptoms via Hamilton Depression Rating Scale (24-item)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Arean, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Weill-Cornell Medical Center, White Plains, New York
  - University of Washington Department of Psychiatry and Behavioral Sciences, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will make de-identified data available to all parties interested.